CLINICAL TRIAL: NCT07344246
Title: Efficacy and Safety of Systemic Dexamethasone Palmitate Treatments in Acute and Subacute Herpes Zoster Pain：a Randomized, Prospective, Multicenter, Blinded Endpoint, Open-label Controlled Trial
Brief Title: Efficacy and Safety of Intravenous Dexamethasone Palmitate Treatments in Acute and Subacute Herpes Zoster Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-440-02
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Herpes Zoster Pain
MeSH Terms: interventions — Injections, Intramuscular; Infusions, Intravenous; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intramuscular injection group (IM group) (Experimental): patients were allocated to receive the same standard antiviral therapy as the control group. Additionally, after routine physical examinations and vital sign monitor, they received 8 mg dexamethasone palmitate administered via intramuscular injection (IM group)
  Interventions: Drug: intramuscular injection (IM group) or intravenous infusion (IV group)
- intravenous infusion group (IV group) (Experimental): patients were allocated to receive the same standard antiviral therapy as the control group. Additionally, after routine physical examinations and vital sign monitor, they received 8 mg dexamethasone palmitate administered via intravenous infusion
  Interventions: Drug: intramuscular injection (IM group) or intravenous infusion (IV group)
- control group (No Intervention): HZ patients with onset of skin lesions within 72 hours received a standard seven-day course antiviral therapy with famciclovir 500 mg three times daily. Besides, they received daily 300 mg pregabalin in divided doses (150 mg/12 hours). Once the patient report mild pain (VAS ≤ 3), the trial for reducing the pregabalin dose was done. If the VAS value increased to more than 3, the patient was returned to the last controllable pregabalin dose. Furthermore, nonsteroidal anti-inflammatory drug celecoxib (200 mg on request, up to two times daily) and tramadol (100 mg on request, up to 400mg daily) will be available for as-needed analgesia, so that a sufficient pain therapy is guaranteed.

INTERVENTIONS:
Drug: intramuscular injection (IM group) or intravenous infusion (IV group) — after routine physical examinations and vital sign monitor, they received 8 mg dexamethasone palmitate administered via intramuscular injection (IM group) or intravenous infusion (IV group)
  Arms: intramuscular injection group (IM group); intravenous infusion group (IV group)

SUMMARY:
This is a randomized, prospective, multicenter, open-label, blinded-endpoint study investigating the efficacy and safety of dexamethasone palmitate (DXP) for treating acute and subacute herpes zoster (shingles) pain.

The study consists of four parallel sub-studies, each designed to answer a specific question:

Study 1: Compares intramuscular (IM) vs. intravenous (IV) administration of DXP (8mg) against standard therapy alone.

Study 2: Compares two different IV doses of DXP (4mg vs. 8mg) against standard therapy.

Study 3: For HZ on the body trunk, compares IM injection vs. tender point infiltration vs. paravertebral nerve block (all containing 8mg DXP).

Study 4: For HZ on the face (trigeminal nerve), compares IM injection vs. tender point infiltration vs. trigeminal nerve block (all containing 8mg DXP).

Approximately 558 adult patients with HZ rash onset within 90 days and significant pain (VAS ≥7) will be enrolled across the studies. All patients receive standard background therapy, including antiviral medication (famciclovir), pregabalin, and rescue analgesics.

The primary outcome is the change in pain intensity (Visual Analogue Scale, VAS) over 6 months. Secondary outcomes include the incidence of postherpetic neuralgia (PHN) at 3 and 6 months, consumption of pain medications, patient satisfaction, quality of life, and safety.

The goal is to determine if DXP, through its targeted anti-inflammatory action, provides superior pain relief and PHN prevention compared to standard care, with a favorable safety profile across different administration routes.

DETAILED DESCRIPTION:
Herpes zoster (HZ), commonly known as shingles, is a painful condition caused by the reactivation of the varicella-zoster virus (VZV). It typically presents as a unilateral, dermatomal vesicular rash accompanied by severe pain descriptors such as burning, prickling, and electric shock-like sensations. The global incidence of HZ ranges from 2 to 5 per 1000 person-years, with a sharp increase to 5.77-9.85 per 1000 person-years after the age of 50, representing a significant public health burden.

The pain associated with HZ, termed Zoster-Associated Pain (ZAP), progresses through distinct phases: the prodromal phase (1-5 days before rash), the acute phase (≤30 days after rash onset), and the subacute phase (31-89 days after rash onset). The most debilitating complication is Postherpetic Neuralgia (PHN), defined as pain persisting for 90 days or more after rash onset. PHN affects approximately 30% of HZ patients and can persist for years, severely diminishing quality of life. A cornerstone of HZ management is the early and aggressive treatment of acute and subacute ZAP to achieve symptomatic relief and potentially prevent the transition to the chronic neuropathic pain state of PHN.

The pathophysiology of ZAP evolves over time. Acute ZAP is predominantly nociceptive, driven by viral replication-induced inflammation, hemorrhagic necrosis of dorsal root ganglia, and tissue edema causing nerve compression. As the disease progresses, peripheral and central sensitization occur, leading to neuropathic pain. Current European guidelines recommend initiating antiviral therapy (e.g., famciclovir) within 72 hours of rash onset to limit viral replication. Pharmacological management of pain typically includes non-opioid analgesics (e.g., NSAIDs like celecoxib), opioid analgesics (e.g., tramadol), and analgesic adjuncts like gabapentin or pregabalin. However, these conventional therapies have limitations, including side effects (gastrointestinal, neuropsychiatric, renal, hepatic) and a limited impact on preventing PHN.

The role of corticosteroids in HZ management remains controversial. Given that inflammation is a key driver of acute pain and neural damage, corticosteroids' potent anti-inflammatory properties are theoretically beneficial. A meta-analysis of systemic corticosteroids (e.g., prednisone) showed efficacy in relieving acute pain but no significant effect on PHN prevention. Furthermore, systemic corticosteroids are associated with well-documented risks, including hyperglycemia, hypertension, weight gain, and gastrointestinal issues. Consequently, current evidence does not support the routine use of systemic corticosteroids for ZAP due to an uncertain risk-benefit profile.

Dexamethasone Palmitate (DXP) is a lipophilic prodrug of dexamethasone with unique pharmacological properties. It has a long biological half-life (36-72 hours) and high lipid solubility. This allows it to be preferentially taken up by phagocytic cells and targeted to sites of inflammation, leading to higher local concentrations and potentially reduced systemic exposure compared to traditional corticosteroids. This targeted action may translate into enhanced efficacy and a more favorable safety profile. Previous studies have explored the use of DXP in local nerve blocks for ZAP, demonstrating promise. However, these procedures are technically demanding, require ultrasound guidance, and carry risks of tissue injury, limiting their widespread applicability.

This study aims to address a critical evidence gap by investigating the efficacy and safety of systemically administered DXP (intramuscular and intravenous) as a more accessible alternative to complex nerve blocks. Furthermore, it will directly compare systemic administration with localized techniques (tender point infiltration, paravertebral, and trigeminal nerve blocks) across different patient populations (spinal and trigeminal nerve HZ) and doses. The overarching hypothesis is that DXP, by effectively controlling early inflammation through various administration routes, will provide superior pain relief and reduce the incidence of PHN compared to standard therapy alone, with an acceptable safety profile.

1.2. Objective

The primary objective of this series of studies is to evaluate the efficacy of different administration routes and doses of Dexamethasone Palmitate (DXP), in combination with standard therapy, versus standard therapy alone, in reducing pain intensity in patients with acute and subacute Herpes Zoster.

The study consists of four distinct but parallel sub-studies:

Study 1: To compare the efficacy of systemic DXP administration (Intramuscular vs. Intravenous injection) against a control group receiving standard therapy.

Study 2: To compare the efficacy of two different intravenous doses of DXP (4 mg vs. 8 mg) against a control group.

Study 3: To compare the efficacy of different injection techniques (Intramuscular vs. Tender Point Infiltration vs. Paravertebral Injection) for HZ affecting spinal nerves (trunk).

Study 4: To compare the efficacy of different injection techniques (Intramuscular vs. Tender Point Infiltration vs. Trigeminal Nerve Block) for HZ affecting the trigeminal nerve (face).

Secondary objectives include:

To compare the incidence of Postherpetic Neuralgia (PHN) at 3 and 6 months post-treatment among the intervention groups.

To assess the consumption of rescue analgesics (celecoxib, tramadol) over time.

To evaluate the consumption of pregabalin over time.

To assess patient satisfaction with the treatment.

To evaluate changes in health-related quality of life (HRQoL).

To monitor and compare the safety and tolerability profiles of all intervention strategies.

1.3. Study Design

Overall Design: This is a prospective, randomized, multicenter, open-label, controlled trial with a blinded endpoint assessment (PROBE design). The trial comprises four independent sub-studies, each with a parallel-group design.

Key Design Features:

Randomization: Participants will be randomly assigned to their respective study groups using a computer-generated random number sequence created with Statistical Package for the Social Sciences (SPSS) version 25.0. Randomization will be stratified by study center to ensure balance across groups for factors like disease duration, baseline pain intensity, and affected dermatome. The allocation ratio is 1:1:1 in all four sub-studies.

Blinding (Masking): This is an open-label study for the treating physicians and patients due to the obvious differences between systemic injections and local procedures. However, to minimize assessment bias, the endpoint is blinded. Specifically, the physicians responsible for post-treatment evaluations during follow-up, the outcome assessors, and the data analysts will be blinded to the treatment group assignments. The operators performing the injections are not involved in any follow-up assessments or data analysis.

Duration: The intervention is a single administration (or a short series for some local techniques). The total study duration for each participant will be approximately 6 months, involving follow-up assessments at Week 1, Week 2, Month 1, Month 3, and Month 6.

Sub-Study Structures:

Study 1 (Systemic Route Comparison):

Group 1: Control Group (n=59): Standard antiviral therapy + Pregabalin + Rescue analgesics.

Group 2: IM Group (n=59): Standard antiviral therapy + Single IM injection of DXP 8 mg + Pregabalin + Rescue analgesics.

Group 3: IV Group (n=59): Standard antiviral therapy + Single IV infusion of DXP 8 mg + Pregabalin + Rescue analgesics.

Study 2 (Intravenous Dose Comparison):

Group 1: Control Group (n=44): Standard antiviral therapy + Pregabalin + Rescue analgesics.

Group 2: 4mg Group (n=44): Standard antiviral therapy + Single IV infusion of DXP 4 mg + Pregabalin + Rescue analgesics.

Group 3: 8mg Group (n=44): Standard antiviral therapy + Single IV infusion of DXP 8 mg + Pregabalin + Rescue analgesics.

Study 3 (Spinal Nerve HZ - Injection Techniques):

Group 1: IM Group (n=43): Standard antiviral therapy + Single IM injection of DXP 8 mg + Pregabalin + Rescue analgesics.

Group 2: TPI Group (n=43): Standard antiviral therapy + Tender Point Infiltration with DXP 8 mg + 1% Lidocaine + Pregabalin + Rescue analgesics.

Group 3: PI Group (n=43): Standard antiviral therapy + Paravertebral Nerve Block with DXP 8 mg + 1% Lidocaine + Pregabalin + Rescue analgesics.

Study 4 (Trigeminal Nerve HZ - Injection Techniques):

Group 1: IM Group (n=40): Standard antiviral therapy + Single IM injection of DXP 8 mg + Pregabalin + Rescue analgesics.

Group 2: TPI Group (n=40): Standard antiviral therapy + Tender Point Infiltration with DXP 8 mg + 1% Lidocaine + Pregabalin + Rescue analgesics.

Group 3: TNI Group (n=40): Standard antiviral therapy + Trigeminal Nerve Block with DXP 8 mg + 1% Lidocaine + Pregabalin + Rescue analgesics.

1.4. Participants (Subject Population)

1.4.1. Eligibility Criteria

Inclusion Criteria (Common to All Studies):

Male or female patients aged 18 to 75 years (inclusive).

Clinical diagnosis of acute or subacute Herpes Zoster, with the onset of the characteristic rash within 90 days prior to enrollment.

Presence of moderate to severe pain, defined as a score of ≥ 7 cm on a 10 cm Visual Analogue Scale (VAS), where 0 represents "no pain" and 10 represents "unbearable pain."

Willing and able to provide written informed consent.

Additional for Study 3: HZ must affect the spinal nerves (cervical, thoracic, or lumbar dermatomes) and the patient must have a tender point count > 4.

Additional for Study 4: HZ must affect the trigeminal nerve (ophthalmic, maxillary, or mandibular branches) and the patient must have a tender point count > 4.

Exclusion Criteria:

Poor general medical condition that, in the investigator's opinion, precludes safe participation in the study or receipt of the assigned intervention.

Known history of substance abuse or narcotic dependence.

Inability to comply with the study protocol, including completion of patient diaries and self-evaluation questionnaires.

Pregnant or lactating women.

Concurrent use of immunosuppressant medications.

Presence of severe, uncontrolled systemic diseases, such as hematological malignancies, active cancers, or significant autoimmune disorders.

Additional for Studies 3 and 4: Presence of a local skin infection at the proposed puncture site for injections/infiltrations.

1.4.2. Sample Size Calculation

Sample size calculations were performed for each sub-study based on preliminary data using Analysis of Variance (ANOVA) with a power of 90% (β=0.1) and a two-sided alpha level of 5% (α=0.05). The calculations accounted for an estimated 10% dropout rate.

Study 1: Based on expected VAS scores at 1 month of 3.8 (Control), 1.5 (IV), and 1.6 (IM), the calculated sample size was 53 per group. Inflating for dropouts, the target enrollment is 59 patients per group (Total N=177).

Study 2: Based on expected VAS scores of 4.2 (Control), 1.7 (4mg IV), and 1.9 (8mg IV), the calculated sample size was 39 per group. Inflating for dropouts, the target enrollment is 44 patients per group (Total N=132).

Study 3: Based on expected VAS scores of 2.2 (TPI), 2.4 (IM), and 3.0 (PI), the calculated sample size was 38 per group. Inflating for dropouts, the target enrollment is 43 patients per group (Total N=129).

Study 4: Based on expected VAS scores of 2.2 (TPI), 2.1 (IM), and 3.4 (TNI), the calculated sample size was 35 per group. Inflating for dropouts, the target enrollment is 40 patients per group (Total N=120).

The total planned enrollment across all four sub-studies is 558 patients.

1.5. Interventions

All patients, regardless of group assignment, will receive a foundation of standard care:

Antiviral Therapy: Famciclovir 500 mg, taken orally three times daily for a 7-day course. This is initiated as early as possible, ideally within 72 hours of rash onset.

Standard Analgesic Regimen:

Pregabalin: A fixed dose of 300 mg daily, administered in divided doses (150 mg every 12 hours). A predefined dose-reduction protocol will be implemented: once a patient reports mild pain (VAS ≤ 3), an attempt to reduce the pregabalin dose will be made. If the VAS increases to >3, the dose will be returned to the last effective level.

Rescue Analgesics:

Celecoxib: 200 mg orally, on an as-needed basis, up to a maximum of two times per day.

Tramadol: 100 mg orally, on an as-needed basis, up to a maximum daily dose of 400 mg.

Prohibited Medications/Therapies: The use of any other oral analgesics is prohibited. Patients are instructed not to undergo any other interventional therapies for their ZAP (e.g., nerve blocks, pulsed radiofrequency) during the study follow-up period.

Study-Specific Interventions:

Control Groups (Studies 1 & 2): Receive only the standard care described above.

Dexamethasone Palmitate (DXP) Interventions:

Systemic Administration (Studies 1 & 2): After routine physical examination and vital sign monitoring, a single dose of DXP will be administered.

IM Injection: Deep intramuscular injection.

IV Infusion: Intravenous infusion over a standardized period.

Local Administration (Studies 3 & 4): Performed by trained clinicians.

Tender Point Infiltration (TPI): Infiltration of the most painful points in the affected dermatome with a solution containing 8 mg DXP and 1% lidocaine.

Paravertebral Injection (PI) / Trigeminal Nerve Block (TNI): A targeted nerve block procedure performed with a solution containing 8 mg DXP and 1% lidocaine.

Post-Intervention Monitoring: Following any injection/infusion, patients will be observed for 30 minutes. If vital signs remain stable, they will be discharged.

1.6. Outcome Measures

1.6.1. Primary Outcome Measure:

Pain Intensity: Change from baseline in pain intensity as measured by the Visual Analogue Scale (VAS, 0-10 cm) at follow-up time points: Week 1, Week 2, Month 1, Month 3, and Month 6.

1.6.2. Secondary Outcome Measures:

Incidence of Postherpetic Neuralgia (PHN): Defined as a VAS score > 0 at 90 days or more after the onset of the HZ rash. Assessed at Month 3 and Month 6.

Rescue Analgesic Consumption: The percentage of patients using rescue analgesics (celecoxib, tramadol) and the average consumption will be recorded at each follow-up (Week 1, 2, Month 1, 3, 6).

Pregabalin Consumption: The mean daily dose of pregabalin will be calculated and compared across groups at each follow-up time point.

Patient Satisfaction: Assessed using a 5-point Likert scale (1=Very Dissatisfied to 5=Very Satisfied) at each follow-up.

Quality of Life (QoL): Evaluated using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire at baseline and each follow-up visit.

Safety and Tolerability:

Incidence and severity of Adverse Events (AEs), particularly those related to corticosteroids (e.g., hyperglycemia, weight gain, hypertension, edema, gastrointestinal symptoms) and procedural complications (e.g., puncture site infection, hematoma, nerve injury, delayed lesion healing).

All AEs will be monitored throughout the study, from the time of informed consent until the final follow-up visit.

1.7. Data Collection and Management

Baseline Data: Demographic and clinical characteristics will be collected at enrollment, including age, gender, BMI, disease duration, affected dermatome, underlying diseases, baseline VAS, and WHOQOL-BREF scores.

Patient Diaries: Patients will be provided with diaries to record daily maximum pain VAS scores, details of all analgesic medications taken (type, dose, time), and any adverse events.

Follow-up Visits: Data will be collected during regular outpatient visits supplemented by structured telephone follow-ups at the specified time points. A designated pain physician at each center will be responsible for data collection and review.

1.8. Statistical Analysis Plan

Statistical analyses will be performed using SPSS version 25.0. The principles of both Intention-to-Treat (ITT) and Per-Protocol (PP) analyses will be applied.

Descriptive Statistics: Continuous variables will be presented as mean ± standard deviation (SD) if normally distributed, or median and interquartile range (IQR) if skewed. Normality will be assessed using the Kolmogorov-Smirnov test. Categorical variables will be expressed as frequencies and percentages.

Between-Group Comparisons:

For continuous, normally distributed data: Independent t-test or ANOVA.

For continuous, skewed data: Mann-Whitney U test or Kruskal-Wallis test.

For categorical data: Chi-square test or Fisher's exact test.

Primary Outcome Analysis: To account for repeated measures and potential confounding factors, the primary analysis for VAS scores over time will use a Repeated-Measures Analysis of Covariance (ANCOVA), adjusting for baseline VAS scores, disease duration, dermatomal level, and other relevant covariates.

Secondary Outcome Analysis:

PHN incidence (binary outcome) will be analyzed using multivariate logistic regression, adjusting for covariates.

Other secondary outcomes (analgesic consumption, QoL) will be analyzed using appropriate parametric or non-parametric tests, with ANCOVA used for continuous outcomes adjusting for baseline values.

Safety Analysis: All safety analyses will be conducted on the Safety Population. The incidence of AEs will be summarized by group.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with onset of HZ rash less than 90 days. 2. HZ affected the trigeminal nerves (ophthalmic/ maxillary/ mandibular nerve). 3. Aged 18 to 75 years (inclusive). 4. Pain intensity ≥ 7 cm on a visual analogue scale (VAS) with 0= 'no pain' to 10='unbearable pain'.

5. Tender point count > 4. 6. Agreed to sign the informed consent form.

Exclusion Criteria:

1. Infection at the puncture site.
2. Poor general situation unable to be treated.
3. A history of abuse of narcotics.
4. Non-compliance or inability to complete the self-evaluation questionnaires.
5. Pregnancy or lactation.
6. Patients using immunosuppressants and those with severe systemic diseases such as hematological malignancies, cancers, or autoimmune disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 954 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS scores at different follow-up time points. | week 1, week 2, month 1, month 3, month 6
  VAS scores at week 1, week 2, month 1, month 3, month 6 following the treatments.

SECONDARY OUTCOMES:
PHN incidence | month 3 and month 6
  PHN incidence at month 3 and month 6: PHN was defined as VAS >0 for more than 90 days after HZ rash onset

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Study Chair — Beijing Tiantan Hospital, Capital Medical University,Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article will be shared following publication. The data will be available with researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be directed to the corresponding author. Data requestors will need to sign a data access agreement to gain access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified IPD and supporting documents will become available starting 6 months after the publication of the primary trial results . The data will be accessible for a period of 5 years This timeframe aligns with standard data sharing policies to ensure data are available while the research remains relevant.
Access Criteria: Who can access the IPD: Qualified researchers with a sound scientific proposal.
  What data will be accessible: De-identified individual participant data and the study protocol.
  How to access it: Proposals should be submitted to the corresponding author. Approved requestors will need to sign a data access agreement before gaining access via a secure file-sharing service.